CLINICAL TRIAL: NCT01230502
Title: Donor Specific Regulation (DSR) Guided Tacrolimus Withdrawal to Myfortic Monotherapy in Liver Transplantation
Brief Title: Mycophenolic Acid (MPA) Monotherapy in Liver Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient study population to meet study objective
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW H-2010-0121; CERL080AUS80T (Other Grant/Funding Number: Novartis Pharmaceuticals)
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Liver Transplant
Keywords: immunosuppression; anti-rejection; immune tolerance
MeSH Terms: interventions — Mycophenolic Acid; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 3: Donor Specific Regulation (DSR) -, standard of care (Active Comparator): Subjects who test Donor Specific Regulation (DSR) negative will not be randomized to possible tacrolimus withdrawal, and will remain on standard of care immunosuppression.
  Interventions: Other: data and sample collection
- Group 2 Donor Specific Regulation (DSR) +; standard of care (Active Comparator): Subjects that are Donor Specific Regulation (DSR) positive and randomized (1:1) to Group 2 will remain on standard of care immunosuppression.
  Interventions: Other: data and sample collection
- Group 1 Donor Specific Regulation (DSR) +, MPA monotherapy (Experimental): Group 1 Donor Specific Regulation (DSR) +, Mycophenolic acid (MPA) monotherapy:
  Subjects that are Donor Specific Regulation (DSR) positive and randomized (1:1) to Group 1 will begin a taper off tacrolimus for 6 months, after repeat DSR testing at 6 months subject will either discontinue tacrolimus if they remain DSR negative or remain at reduced dose if converted to DSR positive
  Interventions: Drug: Group 1 Donor Specific Regulation (DSR) +, Mycophenolic acid (MPA) monotherapy

INTERVENTIONS:
Drug: Group 1 Donor Specific Regulation (DSR) +, Mycophenolic acid (MPA) monotherapy — Group 1 Donor Specific Regulation (DSR) +, MPA monotherapy
  Mycophenolate sodium : Myfortic therapy will be maintained at a target dose of 720mg BID.
  Tacrolimus doses will be lowered to achieve levels of 3-5 ng/ml. 6 months later, immunological monitoring will be repeated and tacrolimus will be completely discontinued if the subject remains DSR + without development of donor specific antibodies (DSA). Those who become DSR- or develop DSA will remain on a tacrolimus dose achieving levels of 3-5 ng/ml, and will not undergone any additional reduction.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples.
  Other Names: Myfortic
  Arms: Group 1 Donor Specific Regulation (DSR) +, MPA monotherapy
Other: data and sample collection — Group 2 : Donor specific regulation (DSR) + standard of care:
  These subjects will be maintained on standard of care immunosuppression consisting of Tacrolimus and Mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples
  Arms: Group 2 Donor Specific Regulation (DSR) +; standard of care
Other: data and sample collection — Group 3 : Donor specific regulation (DSR) - standard of care:
  These subjects are those who were DSR negative and/or DSA positive at enrollment and therefore are not eligible for the withdrawal aspect of the study. These subjects will be maintained on standard of care immunosuppression consisting of Tacrolimus and Mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment. These subjects will be asked to provide heath information and donate blood, exclusively for research testing, at the same 6 month intervals as those in the other two arms of the study, and will be followed for 24 months.
  Arms: Group 3: Donor Specific Regulation (DSR) -, standard of care

SUMMARY:
To determine whether long-term maintenance therapy with a single drug (Myfortic) applied using advanced immunologic monitoring tools in selected patients can lead to superior native kidney function at 2 years without resulting in increased acute rejection episodes or deterioration of liver allograft function.

DETAILED DESCRIPTION:
The hypothesis to be tested is that donor-microchimerism in specific cell populations promotes the development of donor-specific regulation which in turn allows for long-term maintenance therapy with a single drug (Myfortic) in selected patients leading to superior long-term outcomes. Subjects will be enrolled post-transplantation and will be liver transplant recipients who meet the eligibility and exclusion criteria. We will use post-transplant monitoring for donor-specific immunologic regulation (DSR+/ DSA negative) to direct the withdrawal of patients to Myfortic monotherapy. Donor microchimerism, DSR, DSA development will be performed on samples obtained every six months from patients on study. The ultimate objective of the study is to use immunologic monitoring to develop a rational approach to achieving individualized immunosuppression for liver transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ages 18 years and older who have received a primary liver transplant from a deceased donor for end stage liver disease *(ESLD).
* Women of child-bearing potential must have a negative serum pregnancy test at the time of screening and agree to use a medically acceptable method of contraception throughout the study and for 3 months following discontinuation of study treatment.

Exclusion Criteria:

* Recipients of multi-organ transplants.
* Recipients with positive crossmatch with their donor (current or previously).
* Subjects with a screening white blood cell count ≤ 2,000 mm3 or absolute neutrophil count (ANC) ≤ 1000, platelet count ≤ 100,000 mm3.
* Recipients with a hematocrit < 32.
* History of malignancy within 5 years of enrollment (except for adequately treated basal cell or squamous cell carcinoma of the skin).
* Subjects who are positive for hepatitis C, hepatitis B surface antigen, or HIV.
* Subjects with previous intolerance to full dose MPA agent.
* Subjects with a history of acute rejection within 6 months prior to study enrollment.
* Subjects who have had chronic ductopenic rejection.
* Subjects who had rejection in the first-year post-transplant and are less than 3 years post-transplant.
* Subjects who had rejection requiring treatment with thymoglobulin or Orthoclone-OKT3 (OKT3) at anytime post-transplant.
* Original cause of ESLD related to autoimmune diseases such as autoimmune hepatitis, primary biliary cirrhosis, and primary sclerosing cholangitis.
* Subjects who have received an investigational drug within 4 weeks of study entry.
* Subjects with a history of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Female subjects who are pregnant or nursing or females who are unwilling to use contraception during the study.
* Subjects who are currently receiving any therapy for immunosuppression other than a MPA agent and tacrolimus.
* Subjects with a history of hepatocellular carcinoma (T2 >).
* Subjects with severe coexisting disease or presenting with any unstable medical condition which could affect study objectives.
* Subjects who have a known hypersensitivity to tacrolimus or mycophenolate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Will Burlingham, PhD, Principal Investigator — University of Wisconsin, Madison; Anthony D'Alessandro, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin- Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants consented and were enrolled in the study. However, 2 of the subjects screen failed and did not participate in the study beyond providing their consent to participate. Thus only 9 subjects consented to and "started" the study and these 9 subjects are analyzed in the results.
Groups:
- Group 3: Donor Specific Regulation (DSR) -, Standard of Care: Subjects who test Donor specific regulation (DSR) negative will not be randomized to possible tacrolimus withdrawal, and will remain on standard of care immunosuppression.
  data and sample collection: Group 3 : DSR (-) standard of care:
  These subjects are those who were DSR negative and/or DSA positive at enrollment and therefore are not eligible for the withdrawal aspect of the study. These subjects will be maintained on standard of care immunosuppression consisting of tacrolimus and mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment. These subjects will be asked to provide heath information and donate blood, exclusively for research testing, at the same 6 month intervals as those in the other two arms of the study, and will be followed for 24 months.
- Group 2 Donor Specific Regulation (DSR) +; Standard of Care: Subjects that are DSR (donor specific regulation) positive and randomized (1:1)to Group 2 will remain on standard of care immunosuppression.
  data and sample collection: Group 2 : DSR (+)standard of care:
  These subjects will be maintained on standard of care immunosuppression consisting of Tacrolimus and Mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples
- Group 1 Donor Specific Regulation (DSR) +, MPA Monotherapy: Subjects that are Donor specific regulation (DSR) positive and randomized (1:1) to Group 1 will begin a taper off tacrolimus for 6 months, after repeat DSR testing at 6 months subject will either discontinue tacrolimus if they remain DSR negative or remain at reduced dose if converted to DSR positive
  Withdrawal of Tacrolimus to mycophenolate monotherapy: Group 1:
  Mycophenolate sodium : Myfortic therapy will be maintained at a target dose of 720mg BID.
  Tacrolimus doses will be lowered to achieve levels of 3-5 ng/ml. 6 months later, immunological monitoring will be repeated and tacrolimus will be completely discontinued if the subject remains DSR + without development of donor specific antibodies (DSA). Those who become DSR- or develop DSA will remain on a tacrolimus dose achieving levels of 3-5 ng/ml, and will not undergone any additional reduction.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples.
Period: Overall Study
Arm/Group | Group 3: Donor Specific Regulation (DSR) -, Standard of Care | Group 2 Donor Specific Regulation (DSR) +; Standard of Care | Group 1 Donor Specific Regulation (DSR) +, MPA Monotherapy
Started | 9 | 0 | 0
Completed | 9 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 3: Donor Specific Regulation DSR -, Standard of Care: Subjects who test DSR (donor specific regulation) negative will not be randomized to possible tacrolimus withdrawal, and will remain on standard of care immunosuppression.
  data and sample collection: Group 3 : DSR(-) standard of care:
  These subjects are those who were DSR negative and/or DSA positive at enrollment and therefore are not eligible for the withdrawal aspect of the study. These subjects will be maintained on standard of care immunosuppression consisting of tacrolimus and mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment. These subjects will be asked to provide heath information and donate blood, exclusively for research testing, at the same 6 month intervals as those in the other two arms of the study, and will be followed for 24 months.
- Group 2 Donor Specific Regulation DSR +; Standard of Care: Subjects that are DSR (donor specific regulation) positive and randomized (1:1)to Group 2 will remain on standard of care immunosuppression.
  data and sample collection: Group 2 : DSR(+) standard of care:
  These subjects will be maintained on standard of care immunosuppression consisting of tacrolimus and mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples
- Group 1 Donor Specific Regulation (DSR) +, MPA Monotherapy: Subjects that are DSR (donor specific regulation) positive and randomized (1:1)to Group 1 will begin a taper off tacrolimus for 6 months, after repeat DSR testing at 6 months subject will either discontinue tacrolimus if they remain DSR negative or remain at reduced dose if converted to DSR positive
  Withdrawal of Tacrolimus to mycophenolate monotherapy: Group 1:
  Mycophenolate sodium : Myfortic therapy will be maintained at a target dose of 720mg BID.
  Tacrolimus doses will be lowered to achieve levels of 3-5 ng/ml. 6 months later, immunological monitoring will be repeated and tacrolimus will be completely discontinued if the subject remains DSR + without development of donor specific antibodies (DSA). Those who become DSR- or develop DSA will remain on a tacrolimus dose achieving levels of 3-5 ng/ml, and will not undergone any additional reduction.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples.
- Total: Total of all reporting groups
Arm/Group | Group 3: Donor Specific Regulation DSR -, Standard of Care | Group 2 Donor Specific Regulation DSR +; Standard of Care | Group 1 Donor Specific Regulation (DSR) +, MPA Monotherapy | Total
Number analyzed (Participants) | 9 | 0 | 0 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14.757) |  |  | 51 (14.76)
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 8 |  |  | 8
  >=65 years | 1 |  |  | 1
Gender [Number; unit: participants]
  Female | 3 |  |  | 3
  Male | 6 |  |  | 6
Region of Enrollment [Number; unit: participants]
  United States | 9 |  |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Modification of Diet in Renal Disease (MDRD) Estimation of Glomerular Filtration Rate (GFR)
Description: This outcome measure is used to determine if the reduction of calcineurin inhibitor immunosuppression leads to improved native kidney function. Native kidney function is assessed using the Modification of Diet in Renal Disease (MDRD) estimation of glomerular filtration rate (GFR) from serum or plasma creatinine samples at the reported time points.
  Reference intervals include:
  Healthy 18 years and up: 60-120 mL/min/1.73 sqm Chronic kidney disease: GFR < 60 mL/min/1.73 sqm Kidney failure: GFR < 15 mL/min/1.73 sqm
Time Frame: 6 months post enrollment/randomization
Measure: Mean (Standard Deviation); unit: mL/min/1.73 sqm
Groups:
- Group 3: DSR (-), Standard of Care: Subjects who test DSR negative will not be randomized to possible tacrolimus withdrawal, and will remain on standard of care immunosuppression.
  data and sample collection: Group 3 : DSR (-) standard of care:
  These subjects are those who were DSR negative and/or DSA positive at enrollment and therefore are not eligible for the withdrawal aspect of the study. These subjects will be maintained on standard of care immunosuppression consisting of tacrolimus and mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment. These subjects will be asked to provide heath information and donate blood, exclusively for research testing, at the same 6 month intervals as those in the other two arms of the study, and will be followed for 24 months.
- Group 2 DSR (+); Standard of Care: Subjects that are DSR positive and randomized (1:1)to Group 2 will remain on standard of care immunosuppression.
  data and sample collection: Group 2 : DSR (+)standard of care:
  These subjects will be maintained on standard of care immunosuppression consisting of tacrolimus and mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples
- Group 1 DSR (+), Withdrawal of Tacrolimus to MPA Monotherapy: Subjects that are DSR positive and randomized (1:1)to Group 1 will begin a taper off tacrolimus for 6 months, after repeat DSR testing at 6 months subject will either discontinue tacrolimus if they remain DSR negative or remain at reduced dose if converted to DSR positive
  Withdrawal of Tacrolimus to mycophenolate monotherapy: Group 1:
  Mycophenolate sodium : Myfortic therapy will be maintained at a target dose of 720mg BID.
  Tacrolimus doses will be lowered to achieve levels of 3-5 ng/ml. 6 months later, immunological monitoring will be repeated and tacrolimus will be completely discontinued if the subject remains DSR + without development of donor specific antibodies (DSA). Those who become DSR- or develop DSA will remain on a tacrolimus dose achieving levels of 3-5 ng/ml, and will not undergone any additional reduction.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples.
Arm/Group | Group 3: DSR (-), Standard of Care | Group 2 DSR (+); Standard of Care | Group 1 DSR (+), Withdrawal of Tacrolimus to MPA Monotherapy
Number analyzed (Participants) | 7 | 0 | 0
mL/min/1.73 sqm | 60.14 (16.39) |  |

2. Primary Outcome: Modification of Diet in Renal Disease (MDRD) Estimation of Glomerular Filtration Rate (GFR)
Description: as for outcome 1
Time Frame: 12 months post enrollment/randomization
Measure: Mean (Standard Deviation); unit: mL/min/1.73 sqm
Groups:
- Group 3: Donor Specific Regulation (DSR) -, Standard of Care: Subjects who test DSR negative will not be randomized to possible tacrolimus withdrawal, and will remain on standard of care immunosuppression.
  data and sample collection: Group 3 : DSR (-) standard of care:
  These subjects are those who were DSR negative and/or DSA positive at enrollment and therefore are not eligible for the withdrawal aspect of the study. These subjects will be maintained on standard of care immunosuppression consisting of tacrolimus and mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment. These subjects will be asked to provide heath information and donate blood, exclusively for research testing, at the same 6 month intervals as those in the other two arms of the study, and will be followed for 24 months.
- Group 2 Donor Specific Regulation (DSR) +; Standard of Care: Subjects that are DSR positive and randomized (1:1)to Group 2 will remain on standard of care immunosuppression.
  data and sample collection: Group 2 : DSR (+)standard of care:
  These subjects will be maintained on standard of care immunosuppression consisting of tacrolimus and mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples
- Group 1 Donor Specific Regulation (DSR) +, MPA Monotherapy: Subjects that are DSR positive and randomized (1:1) to Group 1 will begin a taper off tacrolimus for 6 months, after repeat DSR testing at 6 months subject will either discontinue tacrolimus if they remain DSR negative or remain at reduced dose if converted to DSR positive
  Withdrawal of Tacrolimus to mycophenolate monotherapy: Group 1:
  Mycophenolate sodium : Myfortic therapy will be maintained at a target dose of 720mg BID.
  Tacrolimus doses will be lowered to achieve levels of 3-5 ng/ml. 6 months later, immunological monitoring will be repeated and tacrolimus will be completely discontinued if the subject remains DSR + without development of donor specific antibodies (DSA). Those who become DSR- or develop DSA will remain on a tacrolimus dose achieving levels of 3-5 ng/ml, and will not undergone any additional reduction.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples.
Arm/Group | Group 3: Donor Specific Regulation (DSR) -, Standard of Care | Group 2 Donor Specific Regulation (DSR) +; Standard of Care | Group 1 Donor Specific Regulation (DSR) +, MPA Monotherapy
Number analyzed (Participants) | 5 | 0 | 0
mL/min/1.73 sqm | 82.4 (28.34) |  |

ADVERSE EVENTS:
Groups:
- Group 3: DSR (Donor Specific Regulation) (-), Standard of Care: Subjects who test Donor specific regulation (DSR) negative will not be randomized to possible tacrolimus withdrawal, and will remain on standard of care immunosuppression.
  data and sample collection: Group 3 : DSR(-) standard of care:
  These subjects are those who were DSR negative and/or DSA positive at enrollment and therefore are not eligible for the withdrawal aspect of the study. These subjects will be maintained on standard of care immunosuppression consisting of tacrolimus and mycophenolate sodium with no reduction in tacrolimus dose during the 24 months of study enrollment. These subjects will be asked to provide heath information and donate blood, exclusively for research testing, at the same 6 month intervals as those in the other two arms of the study, and will be followed for 24 months.
- Group 2 DSR (Donor Specific Regulation) (+); Standard of Care: Subjects that are Donor specific regulation (DSR) positive and randomized (1:1)to Group 2 will remain on standard of care immunosuppression.
  data and sample collection: Group 2 : DSR(+) standard of care:
  These subjects will be maintained on standard of care immunosuppression consisting of tacrolimus and mycophenolate sodium (MPS) with no reduction in tacrolimus dose during the 24 months of study enrollment.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples
- Group 1 DSR (Donor Specific Regulation) (+),MPA Monotherapy: Subjects that are Donor specific regulation DSR positive and randomized (1:1) to Group 1 will begin a taper off tacrolimus for 6 months, after repeat DSR testing at 6 months subject will either discontinue tacrolimus if they remain DSR negative or remain at reduced dose if converted to DSR positive
  Withdrawal of Tacrolimus to mycophenolate monotherapy: Group 1:
  Mycophenolate sodium : Myfortic therapy will be maintained at a target dose of 720mg BID.
  Tacrolimus doses will be lowered to achieve levels of 3-5 ng/ml. 6 months later, immunological monitoring will be repeated and tacrolimus will be completely discontinued if the subject remains DSR + without development of donor specific antibodies (DSA). Those who become DSR- or develop DSA will remain on a tacrolimus dose achieving levels of 3-5 ng/ml, and will not undergone any additional reduction.
  Subjects will be followed for 24 months at 6 month intervals, and will provide health information and blood samples.
Arm/Group | Group 3: DSR (Donor Specific Regulation) (-), Standard of Care | Group 2 DSR (Donor Specific Regulation) (+); Standard of Care | Group 1 DSR (Donor Specific Regulation) (+),MPA Monotherapy
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/9 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI, or his designee, must notify the sponsor at least (10) days, if possible, or as soon as possible, prior to submitting this information.